CLINICAL TRIAL: NCT01537757
Title: An Open-Label, Two-Part, Single-Dose Study to Investigate the Pharmacokinetics of MK-8931 in Subjects With Renal Insufficiency (Protocol No. MK-8931-009 [P08535])
Brief Title: A Two-Part, Single-Dose Study of the Pharmacokinetics of MK-8931 in Subjects With Renal Insufficiency (MK-8931-009 [P08535])
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08535; MK-8931-009 (Other: Schering -Plough)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — verubecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1, Panel A - Severe Renal Impairment Group (Experimental)
  Interventions: Drug: MK-8931
- Part 1, Panel B - Healthy Control Group to Match Panel A (Experimental)
  Interventions: Drug: MK-8931
- Part 2, Panel C - Moderate Renal Impairment Group (Experimental)
  Interventions: Drug: MK-8931
- Part 2, Panel D - Healthy Control Group to Match Panel C (Experimental)
  Interventions: Drug: MK-8931
- Part 2, Panel E - Mild Renal Impairment Group (Experimental)
  Interventions: Drug: MK-8931
- Part 2, Panel F - Healthy Control Group to Match Panel E (Experimental)
  Interventions: Drug: MK-8931

INTERVENTIONS:
Drug: MK-8931 — Single dose, administered as oral capsules

SUMMARY:
This study will assess the pharmacokinetics of MK-8931, a ß-secretase inhibitor, in participants with renal insufficiency. In Part 1 of the study, pharmacokinetics of MK-8931 in participants with severe renal disease and in healthy matched control participants will be studied. If data from Part 1 confirms that severe renal impairment does not alter the pharmacokinetics of MK-8931 to the extent requiring dosage adjustment, then no further study will be required and Part 2 will be optional. If the data does not support this conclusion, then Part 2 will be conducted to study the pharmacokinetics of MK-8931 in participants with moderate and mild renal impairment compared to healthy matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≤39 kg/m^2
* No clinically significant abnormality on electrocardiogram
* Female participant must be postmenopausal or surgically sterilized
* Non-vasectomized men must agree to use a condom with spermicide or abstain from sexual intercourse, during the trial and for 3 months after stopping the medication

Inclusion Criteria Specific to Renally Impaired Participants:

* Clinical diagnosis of renal insufficiency based on Estimated Glomerular Filtration rate (eGFR): severely decreased eGFR, defined as <30 mL/min/1.73m^2 and participant is not on dialysis; moderately decreased eGFR, defined as ≥30 to <60 mL/min/1.73m^2; mildly decreased eGFR, defined as ≥60 to <80 mL/min/1.73m^2
* Stable baseline health based on medical history, physical examination, vital signs, and laboratory tests

Inclusion Criterion Specific to Healthy Participants:

* eGFR ≥80 mL/min/1.73m^2

Exclusion Criteria:

* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug, including history or presence of inflammatory bowel disease, gastrointestinal or rectal bleeding; presence of active ulcer; history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; history of pancreatic injury or pancreatitis; history or presence of liver disease or liver injury; history of urinary obstruction or difficulty in voiding
* History of any infectious disease within 4 weeks prior to drug administration
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCV) or human immunodeficiency virus (HIV)
* History of risk factors for Torsades de Pointes (e.g., heart failure/cardiomyopathy or family history of Long QT Syndrome)
* Participant has had a kidney removed or has a functioning renal transplant
* History of alcohol or drug abuse in the past 2 years
* Blood donation or loss of significant volume of blood in the past 60 days prior to dosing
* Previously received MK-8931
* History of significant multiple and/or severe allergies (including latex allergy), or anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* History of malignancy occurring within the 5 years immediately before screening, except for a participant who has been adequately treated for basal cell or squamous cell skin cancer; or in situ cervical cancer; or

localized prostate carcinoma; or has undergone potentially curative therapy with no evidence of recurrence ≥1 year post-therapy

Exclusion Criteria Specific to Renally Impaired Participants:

* Rapidly fluctuating renal function as determined by historical measurements
* Suspected renal artery stenosis

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of MK-8931 | Predose through 120 hours post single dose of MK-8931

SECONDARY OUTCOMES:
Renal clearance (CLr) of MK-8931 | Predose through 120 hours post single dose of MK-8931
Fraction of MK-8931 dose excreted in urine (fe) | Predose through 120 hours post single dose of MK-8931